CLINICAL TRIAL: NCT00215397
Title: Study in Patients With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Director, Clinical Affairs, Dey
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DL-053
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2008-02

CONDITIONS: Asthma
Keywords: Asthma; Formoterol; Fumarate
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate

INTERVENTIONS:
Drug: Formoterol Fumarate

SUMMARY:
The purpose of this study is to determine which dose of the investigational drug is the most safe and effective in the treatment of asthma compared to the control drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of asthma

Exclusion Criteria:

* Current asthma exacerbation or recent asthma exacerbation, requiring hospitalization
* History of smoking
* Debilitating systemic and/or life-threatening diseases.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16
Dates: Primary Completion 2003-02 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable is the measure of lung function.

SECONDARY OUTCOMES:
Secondary outcomes include change in lung function, as well as in vital signs.
Physical exams, AE reporting, etc.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Site, Long Beach, California
  - Research Site, Denver, Colorado
  - Research Site, Medford, Oregon